CLINICAL TRIAL: NCT04967157
Title: A Randomized, Parallel, Double-Blind, Placebo-Controlled Study to Assess the Cognitive Effects of a Citicoline Supplement (Cognizin®) on Attention in Healthy Men and Women
Brief Title: Cognitive Effects of Citicoline on Attention in Healthy Mean and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirin Holdings Company, Limited (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIO-2104
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Intervention: Dietary Supplement: Placebo supplement
  Interventions: Dietary Supplement: Placebo supplement
- Cognizin® (Experimental): Intervention: Dietary Supplement: Citicoline supplement
  Interventions: Dietary Supplement: Citicoline supplement

INTERVENTIONS:
Dietary Supplement: Placebo supplement — Cellulose
  Other Names: Placebo
  Arms: Placebo
Dietary Supplement: Citicoline supplement — Cognizin ®
  Other Names: Cognizin ®
  Arms: Cognizin®

SUMMARY:
The objective of this trial is to determine the effects of citicoline on cognitive performance for attention in healrhy Men and Women compared to a placebo.

DETAILED DESCRIPTION:
This study is a 12-week, randomized, double-blind, placebo-controlled trial of citicoline in healthy men and women. Cognitive assessments will be performed to determine whether citicoline administration improves attention, compared to placebo administration.

**Note: This note is to inform you that the Unique Protocol ID BIO-2104 was unintentionally combined with another Unique Protocol ID, K5-24-01-T0060, resulting in history records that should not be considered as part of the BIO-2104's timeline.

This explanation has been added per PRS instructions to ensure compliance and maintain data integrity in alignment with the protocol.

ELIGIBILITY:
Inclusion Criteria:

* male or female, 35-75 years of age
* Scores ≥ 24 on the MMSE, ≤15 on the CESD-R, and scores below the population median (i.e., below 81.25, above 36.8) on the Gradual CPT
* Self-reported poor attention
* no health conditions that would prevent him or her from fulfilling the study requirements on the basis of medical history and routine laboratory test results
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Principal Investigator.

Exclusion Criteria:

* color blindness
* Known allergy or sensitivity to any of the ingredients in the study products and/or any ingredients of the breakfast meal provided
* major medical or neurological illness
* diagnosis of attention deficit hyperactive disorder (ADHD)
* female who is pregnant, planning to be pregnant during the study period
* requiring treatment with a drug which might obscure the action of the study treatment

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Composite score calculated based on scores from the Computerized Mental Performance Assessment System (COMPASS, Northumbria University, Newcastle upon Tyne, UK) that measure cognitive assessment | 12 weeks

SECONDARY OUTCOMES:
Standardized scores on the Computerized Mental Performance Assessment System (COMPASS, Northumbria University, Newcastle upon Tyne, UK) that measure cognitive assessment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kelley, MD, Principal Investigator — Biofortis Clinical Research, Inc. Addison, Illinois, United States, 60101
Locations (1):
- Biofortis Clinical Research, Inc., Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No